CLINICAL TRIAL: NCT02430324
Title: Post Traumatic Cerebral Infarction Increases Mortality and Morbidity in Patients With Moderate or Severe Head Trauma. The Multicenter Italian INCEPT (INfarto CErebrale Post-Traumatico) Study
Brief Title: The Multicenter Italian INCEPT (INfarto CErebrale Post-Traumatico) Study
Status: Completed | Type: Observational
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Collaborators: A.O.U. Città della Salute e della Scienza (Other); Fondazione Poliambulanza Istituto Ospedaliero (Other); A.O. Ospedale Papa Giovanni XXIII (Other); Azienda Ospedaliera San Gerardo di Monza (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other); Azienda Ospedaliero, Universitaria Pisana (Other); Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Dr. Nazzareno Fagoni, Nazzareno Fagoni, MD, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Other Study IDs: prot.1937/2009
Record Dates: First submitted 2015-04-16; First posted 2015-04-30 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: TBI (Traumatic Brain Injury); Stroke Acute
MeSH Terms: conditions — Brain Injuries, Traumatic; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TBI, no cerebral infarction: patients with moderate or severe brain injury that do not develop posttraumatic cerebral infarction
- TBI, posttraumatic cerebral infarction: patients with moderate or severe brain injury that develops posttraumatic cerebral infarction
  Interventions: Other: posttraumatic cerebral infarction

INTERVENTIONS:
Other: posttraumatic cerebral infarction — the difference between groups refers to the developing of cerebral infarction after traumatic brain injury
  Groups: TBI, posttraumatic cerebral infarction

SUMMARY:
Traumatic brain injury (TBI) is a leading cause of death and disability worldwide (Ghajar, 2000). With an estimated annual incidence of up to 500 per 100,000 population and more than 200 hospital admissions per 100,000 admissions in Europe each year, TBI is a major challenge to public health (Lingsma, 2010). Mortality and morbidity after TBI depend on several factors, either associated with patients characteristics, the cause of TBI, the neurological and general severity and secondary brain insults, the structural brain alterations as diagnosed at brain computed tomography (CT) (Rosenfeld, 2012).

The prognostic value of brain CT characteristics is well documented, including the status of basal cisterns, midline shift, the presence and type of intracranial lesions, and traumatic subarachnoid hemorrhage (Maas, 2008). Postraumatic cerebral ischemia, which includes functionally impaired yet still viable tissue, so-called ischemic penumbra, and irreversible cerebral infarction (PTCI), is frequent in patients who die after moderate or severe head trauma (Stocchetti, 2014).

Evidence of antemortem occurrence of PTCI is limited to three single-center retrospective studies, reporting a varying prevalence of 1.9%, 8% and 19.1% (Mirvis, 1990; Marino, 2006; Tawil, 2008). Increased intracranial pressure (ICP), blunt cerebral vascular injury, need for craniotomy and treatment with recombinant activated factor VII, have been demonstrated to be risk factors for PTCI. In one study, PTCI was an independent risk factor for poor outcome after moderate or severe head trauma with a two-fold increase in mortality and severe disability (Marino, 2006).

PTCI can be an important diagnosis in patients with significant TBI for various reasons. First, it might influence long-term outcome. Second, as an outcome that is measurable, and relevant to survival and lifestyle, PTCI could be used as an outcome measure in randomized controlled trials. Third, diagnosis of PTCI could be used as a standard diagnostic reference to validate early surrogate indicators of cerebral ischemia.

The investigators therefore planned a multi-center prospective study to investigate the impact of PTCI on disability at hospital discharge, and on 6-month morbidity and mortality in a population of moderate and severe adult TBI patients. The investigators also evaluated the role of intracranial hypertension, decreased cerebral perfusion pressure, hypotension and other secondary ischemic insults in determining the appearance of PTCI.

ELIGIBILITY:
Inclusion Criteria:

* age >15 years old,
* with moderate or severe head trauma (GCS <14),
* admitted to ICU. Cases were classified as severe head injury (GCS score < 9), or moderate head injury (GCS score from 9 to 13).

All patients recruited were monitored by means of invasive intracranial pressure (ICP), invasive arterial pressure monitoring, peripheral oxygen saturation, in accordance with published international and local guidelines

Exclusion Criteria:

* age <16 years old,
* mild head trauma,
* absence of invasive ICP or invasive arterial pressure monitoring,
* dying patients,
* absence of brain stem reflexes.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with moderate or severe brain injury, monitored with invasive intracranial pressure.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2009-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Oxford Handicap Scale (OHS) | patients will be evaluated at hospital discharge, an expected average of 3 weeks
  The Oxford Handicap Scale evaluates the outcome as follow: 0 no symptoms, 1 minor symptoms, 2 minor handicap, 3 moderate handicap, 4 severe handicap, 5 death.
  Favourable outcome: 0-3; unfavourable outcome: 4-5
Glasgow Outcome Scale (GOS) | the GOS will be performed 6 months after the hospital admission
  The Glasgow Outcome Scale evaluates the outcome as follow: 1 death, 2 vegetative state, 3 severe handicap, 4 moderate handicap, 5 good recovery.
  Favourable outcome: 4-5; unfavourable outcome: 1-3

SECONDARY OUTCOMES:
Hospital and ICU mortality | at the discharge from ICU, an expected average of 3 weeks; and at the discharge from hospital, an expected average of 6 weeks
  This outcome refers to the mortality during ICU stay and hospital stay
Length of ventilation | during ICU stay, an expected average of 3 weeks
  Days of ventilation, how long does it take to weaning from ventilation
Length of ICU and Hospital stay | at the discharge from ICU, an expected average of 3 weeks; and at the discharge from hospital, an expected average of 6 weeks
  How many days the patients whith cerebral infarction and without cerebral infarction have been in ICU, and how many days the patients were in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Latronico, MD, Study Chair — University of Brescia and AO Spedali Civili di Brescia; Nazzareno Fagoni, MD, Principal Investigator — AO Spedali Civili di Brescia
Locations (1):
- Azienda Ospedaliera Spedali Civili di Brescia, Brescia, Brescia, Italy

REFERENCES:
- [Background] Ghajar J. Traumatic brain injury. Lancet. 2000 Sep 9;356(9233):923-9. doi: 10.1016/S0140-6736(00)02689-1. PMID 11036909
- [Background] Marino R, Gasparotti R, Pinelli L, Manzoni D, Gritti P, Mardighian D, Latronico N. Posttraumatic cerebral infarction in patients with moderate or severe head trauma. Neurology. 2006 Oct 10;67(7):1165-71. doi: 10.1212/01.wnl.0000238081.35281.b5. PMID 17030747
- [Background] Maas AI, Stocchetti N, Bullock R. Moderate and severe traumatic brain injury in adults. Lancet Neurol. 2008 Aug;7(8):728-41. doi: 10.1016/S1474-4422(08)70164-9. PMID 18635021
- [Background] Mirvis SE, Wolf AL, Numaguchi Y, Corradino G, Joslyn JN. Posttraumatic cerebral infarction diagnosed by CT: prevalence, origin, and outcome. AJNR Am J Neuroradiol. 1990 Mar-Apr;11(2):355-60. PMID 2107719
- [Background] Tawil I, Stein DM, Mirvis SE, Scalea TM. Posttraumatic cerebral infarction: incidence, outcome, and risk factors. J Trauma. 2008 Apr;64(4):849-53. doi: 10.1097/TA.0b013e318160c08a. PMID 18404047
- [Background] Rosenfeld JV, Maas AI, Bragge P, Morganti-Kossmann MC, Manley GT, Gruen RL. Early management of severe traumatic brain injury. Lancet. 2012 Sep 22;380(9847):1088-98. doi: 10.1016/S0140-6736(12)60864-2. PMID 22998718
- [Background] Lingsma HF, Roozenbeek B, Steyerberg EW, Murray GD, Maas AI. Early prognosis in traumatic brain injury: from prophecies to predictions. Lancet Neurol. 2010 May;9(5):543-54. doi: 10.1016/S1474-4422(10)70065-X. PMID 20398861
- [Background] Stocchetti N, Maas AI. Traumatic intracranial hypertension. N Engl J Med. 2014 May 29;370(22):2121-30. doi: 10.1056/NEJMra1208708. No abstract available. PMID 24869722
- [Derived] Latronico N, Piva S, Fagoni N, Pinelli L, Frigerio M, Tintori D, Berardino M, Bottazzi A, Carnevale L, Casalicchio T, Castioni CA, Cavallo S, Cerasti D, Citerio G, Fontanella M, Galiberti S, Girardini A, Gritti P, Manara O, Maremmani P, Mazzani R, Natalini G, Patassini M, Perna ME, Pesaresi I, Radolovich DK, Saini M, Stefini R, Minelli C, Gasparotti R, Rasulo FA. Impact of a posttraumatic cerebral infarction on outcome in patients with TBI: the Italian multicenter cohort INCEPT study. Crit Care. 2020 Feb 3;24(1):33. doi: 10.1186/s13054-020-2746-5. PMID 32014041